CLINICAL TRIAL: NCT01369771
Title: An Open-label, Phase IV, Pilot Study, to Evaluate Confocal Microscopic Findings of Cornea, Ocular Signs and Symptoms in Patients With OH or OAG Switching From Latanoprost 0.005% to Preservative Free Tafluprost 0.0015% Eye Drops
Brief Title: The Effects of Preservative-free Prostaglandin Eye Drops in Sign and Symptoms on the Eyes of Patients With Glaucoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: FinnMedi Oy (Industry)
Collaborators: Tampere University (Other); The Laboratory and Pharmacy Public Utility of the Pirkanmaa Hospital District (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S001-2010; 2010-021039-14 (EudraCT Number)
Record Dates: First submitted 2010-07-05; First posted 2011-06-09 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Ocular Hypertension; Open-Angle Glaucoma
Keywords: Confocal microscopic findings; Ocular Hypertension; Open-Angle Glaucoma; Preservative-free eye drops
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — tafluprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tafluprost 0.0015% (Experimental): Open, one arm study. Patients who have been using latanoprost 0.005% eye drops (Xalatan®) as their prior medication (at least 6 months) and who fulfil all the inclusion criteria including the specified ocular symptoms and signs, will switch from latanoprost to the assigned preservative-free tafluprost 0.0015% (Taflotan®)eye drops for twelve (12) months.
  Interventions: Drug: Tafluprost 0.0015%

INTERVENTIONS:
Drug: Tafluprost 0.0015% — Eye Drops, Solution. Topical Use. One single-unit dose pipet of 0.3 ml solution including 0.0015 mg/ ml of Tafluprost once daily in the affected eye(s)for 12 months.
  Other Names: Taflotan®; Taflotan sine®; Saflutan®; Saflutan Conserveermiddelvrij®

SUMMARY:
The objective of this study is to investigate corneal confocal microscopic findings, ocular signs and symptoms in patients on treatment with the preserved prostaglandin analogue latanoprost 0.005% eye drops (Xalatan®) and after the switch to preservative-free prostaglandin analog tafluprost 0.0015% eye drops (Taflotan®). Patients who have been using latanoprost as their prior medication (at least 6 months) and who fulfil all the inclusion criteria including the specified ocular symptoms and signs, will switch from latanoprost 0.005% eye drops to the assigned preservative-free tafluprost 0.0015% eye drops for twelve (12) months.

DETAILED DESCRIPTION:
Primary outcome measures:

1. Change from screening in corneal confocal microscopic findings at month 12
2. Change from screening in ocular symptoms upon non-instillation at month 12
3. Change from screening in ocular signs at month 12

   Safety and QoL variables:
4. Descriptive statistics, identification of change(s) from screening

ELIGIBILITY:
Inclusion Criteria:

* Have provided a written informed consent
* Aged 18 years or more
* A diagnosis of ocular hypertension or open-angle glaucoma (either POAG or capsular glaucoma) in one or both eyes, for which the patient has been regularly using latanoprost 0.005% (Xalatan®) for at least six months before Screening (confirmed in anamnesis)
* In the Screening visit evaluation, the presence of:

At least two ocular symptoms considered for the two eyes together (irritation/burning/stinging, foreign body sensation, tearing, itching or dry eye sensation) of at least mild severity (grade ≥ 2) upon non-instillation OR One ocular symptom of at least mild severity (grade ≥ 2) upon non-instillation AND

At least one of the following ocular signs in either eye with prior treatment:

Fluorescein tear break-up time (fBUT): less than 10 seconds

Corneal and conjunctival fluorescein staining:

Corneal fluorescein staining score of at least grade I OR Combined nasal and temporal staining scores of at least grade II Blepharitis: of at least mild severity (grade ≥ 1) Conjunctival redness/hyperemia: of at least mild severity (grade 1) Tear production: 10 mm or less on Schirmer test

* A best corrected ETDRS visual acuity score of +0.6 logMAR or better in both eyes
* Negative pregnancy test result at the screening visit, or, consistently and correctly used reliable method of contraception during the study
* Are willing to follow instructions

Exclusion Criteria:

* Females who are pregnant, nursing or planning a pregnancy, or females of childbearing potential who are not using a reliable method of contraception
* Anterior chamber angle in either eye to be treated less than grade 2 according to Schaffer classification as measured by gonioscopy
* Any corneal abnormality or other condition preventing reliable applanation tonometry, including prior refractive eye surgery
* IOP greater than 22 mmHg at 15:00 IOP measurement in either eye at Screening/Baseline visit
* Use of preserved eye drops (other than latanoprost) including artificial tears at screening or within two weeks prior to screening visit
* Diagnosis of angle-closure glaucoma or secondary glaucoma other than capsular glaucoma in either eye
* Suspected contraindication to tafluprost therapy (hypersensitivity to tafluprost or any of the excipients)
* Glaucoma filtration surgery or any other ocular surgery (including ocular laser procedures) within 6 months prior to Screening in eye(s) to be treated with study medication
* Use of contact lenses at Screening or during the study
* Any ocular (e.g. aphakia, pseudophakia with torn posterior lens capsule2 or anterior chamber lenses,known risk factors for cystoid macular oedema or iritis/uveitis), systemic or psychiatric disease/condition (e.g.uncontrolled arterial hypertension, diabetes) that may put the patient at a significant risk or may confound the study results or may interfere significantly with the patient's participation in the study as judged by the investigator
* Current alcohol or drug abuse
* Current participation in another clinical trial involving an investigational drug/device, or participation in such a trial within the last 30 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from screening in corneal confocal microscopic findings at month 12 | Baseline and Month 12

SECONDARY OUTCOMES:
Change from screening in ocular symptoms and signs upon non-instillation | Baseline and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Hannu Uusitalo, MD, PhD, Principal Investigator — Clinical Trial Center, FinnMedi Oy
Locations (1):
- FinnMedi Oy, Clinical Trial Center, Tampere, Pirkanmaa District, Finland